CLINICAL TRIAL: NCT00742521
Title: Mechanisms of Hypoglycemia Associated Autonomic Dysfunction, Question 3
Brief Title: Mechanisms of Hypoglycemia Associated Autonomic Dysfunction, Q.3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: IRB#010733; HL056693-10
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Type 1 Diabetes
Keywords: cortisol; catecholamines; Type 1 DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Euglycemic glucose clamp procedure x 2 on Day 1 and hypoglycemic glucose clamp procedure on Day 2. Control study
  Interventions: Procedure: glucose clamp
- 2 (Active Comparator): Hypoglycemic glucose clamp procedure x 2 on Day 1 and hypoglycemic glucose clamp procedure on Day 2. Control study
  Interventions: Procedure: glucose clamp
- 3 (Active Comparator): Euglycemic glucose clamp procedure x 2 with cortisol infusion of 2ug/kg on Day 1 and hypoglycemic glucose clamp procedure on Day 2.
  Interventions: Procedure: glucose clamp
- 4 (Active Comparator): Hyperinsulinemic euglycemic glucose clamp procedure x 2 with cortisol infusion at 1 ug/kg on Day 1 and hyperinsulinemic hypoglycemic glucose clamp procedure on Day 2.
  Interventions: Procedure: glucose clamp

INTERVENTIONS:
Procedure: glucose clamp — Day 1 hyperinsulinemic euglycemic glucose clamp procedure x 2 and Day 2 hyperinsulinemic hypoglycemic glucose clamp procedure
  Arms: 1
Procedure: glucose clamp — Hypoglycemic glucose clamp procedure x 2 on Day 1 and hypoglycemic glucose clamp procedure on Day 2. Control study
  Arms: 2
Procedure: glucose clamp — Hyperinsulinemic euglycemic glucose clamp procedure x 2 with cortisol infusion at 2 ug/kg on Day 1 and hyperinsulinemic hypoglycemic glucose clamp procedure on Day 2.
  Arms: 3
Procedure: glucose clamp — Hyperinsulinemic euglycemic glucose clamp procedure x 2 with cortisol infusion at 1 ug/kg on Day 1 and hyperinsulinemic hypoglycemic glucose clamp procedure on Day 2.
  Arms: 4

SUMMARY:
It has been found that in some cases, when a person with Diabetes Mellitus has an episode of low blood sugar,or hypoglycemia, and then later exercises, he or she is vulnerable to another bout of hypoglycemia during that exercise. The purpose of this study is to determine what factors during the previous bout of hypoglycemia might cause another bout of hypoglycemia while exercising later.

DETAILED DESCRIPTION:
The SPECIFIC AIM of the study outlined in this proposal is to determine if hypoglycemia blunts counterregulatory responses during subsequent exercise in Type 1 Diabetes Mellitus due to physiologic increases in plasma cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with Type 1 Diabetes Mellitus will be studied. Subjects recruited will be 18-50 years, with an HBA1c less than 9.5%, who have been diagnosed with diabetes for >5 years, with no clinical evidence of diabetic tissue complications.

Exclusion Criteria:

* Subjects with known prior cardiac events will be excluded from the study. Additional exclusion criteria:

  1. all medical students (Vanderbilt policy)
  2. prior or current history of poor health
  3. abnormal results following blood and physical examination
  4. pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2001-03; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
catecholamine measures | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States